CLINICAL TRIAL: NCT04937803
Title: Safety and Efficacy of Drug-Coated Balloon for De-novo Lesions in Patients With Acute Coronary Syndromes (DCB-ACS): A Prospective, Multi-Center, Randomized-Controlled Clinical Trial
Brief Title: Safety and Efficacy of Drug-Coated Balloon for De-novo Lesions in Patients With Acute Coronary Syndromes (DCB-ACS)
Acronym: DCB-ACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Collaborators: Daqing Oil Field Hospital (Other); Sichuan Provincial People's Hospital (Other); Tianjin People's Hospital (Other); Peking University First Hospital (Other); Beijing Friendship Hospital (Other); The Third Medical Center, Chinese PLA General Hospital (Unknown); Jining Medical University (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); The First Hospital of Jilin University (Other); General Hospital of Taiyuan Iron & Steel Company (Unknown); Tongji Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Second Affiliated Hospital of Zhengzhou University (Other); Sir Run Run Shaw Hospital (Other); Inner Mongolia People's Hospital (Other)
Responsible Party: Principal Investigator, Yu Bo, The Head of cardiology department, The Second Affiliated Hospital of Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPCTP-2020-001
Record Dates: First submitted 2021-06-10; First posted 2021-06-24 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Drug-Coated Balloon; De Novo Stenosis; Acute Coronary Syndromes; ACS; DCB; Clinical Trial; Coronary Artery Disease
Keywords: Drug-Coated Balloon; De-novo Lesions; Acute Coronary Syndromes; DCB-ACS; ACS; DCB; Clinical Trial; Coronary Artery Disease
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-coated balloon group (Experimental): Patients assigned to drug-coated balloon group will receive angioplasty with drug-coated balloon for treatment of lesions.
  Interventions: Device: Drug-coated balloon
- Stent group (Active Comparator): Patients assigned to drug-eluting stent group will receive a Zotarolimus -Eluting Coronary Stent treatment .
  Interventions: Device: Zotarolimus-Eluting Coronary Stent

INTERVENTIONS:
Device: Drug-coated balloon — Drug-coated balloon is a fast-exchange balloon dilatation catheter, used to treat coronary artery stenosis lesions and improve myocardial blood flow.
  Arms: Drug-coated balloon group
Device: Zotarolimus-Eluting Coronary Stent — Zotarolimus-Eluting Coronary Stent is treated for coronary artery stenosis lesions .
  Arms: Stent group

SUMMARY:
The DCB-ACS trial is a prospective, multi-center, non-inferiority, randomized controlled trail. The purpose of this trial is to evaluate the safety and efficacy of drug-coated balloon(DCB) in de novo lesions for acute coronary syndromes (ACS) .

DETAILED DESCRIPTION:
Patients with ACS and indications for percutaneous coronary intervention were randomly assigned (1:1) to receive angioplasty with DCB or implantation of a Zotarolimus-Eluting Coronary Stent(ZES) . Dual anti-platelet therapy was given according to current guidelines. Follow-up was originally scheduled at by telephone or clinical visit at 1 month, 6 months, 12 months, and 24 months after discharge, and coronary angiography and FFR measurements will be carried out at 9 months.The primary objective is to show non-inferiority of DCB versus drug-eluting stent(DES) regarding the functional assessment of target lesion by FFR at 9 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 Years and <80 years;
2. ACS patients eligible for percutaneous coronary intervention;
3. Successful preparation is defined as ≤ 30% residual stenosis with Thrombolysis in Myocardial Infarction (TIMI) Grade III flow and not evidence of type C-F dissection;
4. Vessel diameter from 2.25mm-4.0 mm ;
5. Lesion length ≤ 28 mm;
6. A single culprit lesion or 1 lesion in each of two vessels ;
7. Eligible for enrollment and provide written informed consent.

Exclusion Criteria:

Clinical Exclusion Criteria：

1. Stable angina or asymptomatic myocardial ischemia;
2. Cardiogenic shock or requiring mechanical support for breathing and circulation;
3. Hemodynamically unstable tachyarrhythmia or bradyarrhythmia;
4. Plan to perform cardiac surgery or non-cardiac surgery within 24 months of percutaneous coronary intervention;
5. A history of stroke within 6 months;
6. History of severe renal insufficiency;
7. Life expectancy < 12 months;
8. Pregnant women;
9. Allergies to aspirin, clopidogrel, ticagrelor, heparin, contrast agents, and paclitaxel, patients with systemic lupus erythematosus or other systemic immune diseases;
10. Patients not suitable for enrollment considered by researcher;
11. Currently participating in another trial before reaching the primary endpoint;
12. Inability to provide informed consent. Image Exclusion Criteria

1. Chronic total occlusion (CTO); 2. Left main lesion; 3. Bifurcation lesions treated with double stents; 4. Moderate to severe distortion, angulation or severe calcification lesions; 5. Coronary artery graft stenosis; 6. In-stent restenosis; 7. To be re-hospitalized for the other scheduled PCI treatment; 8. Myocardial bridge at the target lesion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2023-02-18 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Fractional flow reserve (FFR) | 9 months follow-up
  Fractional flow reserve is the ratio of mean coronary pressure distal of the treated lesion to mean aortic pressure during maximum hyperemia.

SECONDARY OUTCOMES:
Target lesion failure（TLF） | 1 month, 6 months, 9 months, 12 months, 24 months follow-up
  A composite endpoint consisting of cardiac death, target vessel-related myocardial infarction, and revascularization of target lesions
Cardiac death | 1 month, 6 months, 9 months, 12 months, 24 months follow-up
Target vessel-related myocardial infarction | 12 months, 24 months follow-up
Revascularization of target lesion revascularization (TLR) | 1 month, 6 months, 9 months, 12 months, 24 months follow-up
All-cause death and myocardial infarction | 1 month, 6 months, 9 months, 12 months, 24 months follow-up
Major bleeding | 1 month, 6 months, 9 months, 12 months, 24 months follow-up
  Defined as Bleeding Academic Research Consortium type 3 to 5
Procedure success | 1 month
  Including device success, lesion success and procedure success
Patient-oriented composite endpoint (PoCE) | 1 month, 6 months, 9 months, 12 months ,24 months follow-up
  A composite of all-cause mortality, myocardial infarction, and any revascularization.
Diameter stenosis(DS%) | 9 months follow-up
  DS% defined as: (1 - minimal luminal diameter /reference vessel diameter) *100%.
Late lumen loss (LLL） | 9 months follow-up
  The difference between the in-segment minimal lumen diameter after the procedure and at angiographic follow-up, as evaluated by quantitative coronary angiography.
Restenosis rate of target lesion | 9 months
  Diameter stenosis %≥50%
Definite and possible thrombotic events | 2 years
Rehospitalized due to angina | 2 years
Stroke | 2 years
  Diagnosed by a neurologist

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, MD,PhD, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (1):
- The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Jeger RV, Farah A, Ohlow MA, Mangner N, Mobius-Winkler S, Leibundgut G, Weilenmann D, Wohrle J, Richter S, Schreiber M, Mahfoud F, Linke A, Stephan FP, Mueller C, Rickenbacher P, Coslovsky M, Gilgen N, Osswald S, Kaiser C, Scheller B; BASKET-SMALL 2 Investigators. Drug-coated balloons for small coronary artery disease (BASKET-SMALL 2): an open-label randomised non-inferiority trial. Lancet. 2018 Sep 8;392(10150):849-856. doi: 10.1016/S0140-6736(18)31719-7. Epub 2018 Aug 28. PMID 30170854
- [Background] Vos NS, Dirksen MT, Vink MA, van Nooijen FC, Amoroso G, Herrman JP, Kiemeneij F, Patterson MS, Slagboom T, van der Schaaf RJ. Safety and feasibility of a PAclitaxel-eluting balloon angioplasty in Primary Percutaneous coronary intervention in Amsterdam (PAPPA): one-year clinical outcome of a pilot study. EuroIntervention. 2014 Sep;10(5):584-90. doi: 10.4244/EIJV10I5A101. PMID 25256200